CLINICAL TRIAL: NCT03632538
Title: Prospective Analysis of Postoperative Occurrence of Acute Kidney Injury (AKI) and Need for Renal Replacement Therapy After Cardiac Surgery With the Help of New Biomarkers.
Brief Title: AKI Cardiosurgery Diagnostic Study (AKI-CDS)
Acronym: AKI-CDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Dr. Martin Sauer, MD, Principal Investigator, PD Dr. med. habil., University of Rostock
Other Study IDs: A 2018-0092
Record Dates: First submitted 2018-07-27; First posted 2018-08-15 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Acute Kidney Injury; Renal Replacement Therapy
Keywords: Acute Kidney Injury; Cardiac Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Each 8 ml blood drawn from patients for measurement of biomarkes to 6 time points.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male: 20 male adult patients after cardiac surgery. Drawing of patients blood for measurement of biomarkers ("penKid", adrenomedulin, C-terminal alpha-1 antitrypsin peptide) for AKI before and after cardiac surgery (times: 0, 6, 24, 72, 168 hours).
  Interventions: Diagnostic Test: Biomarker ("penKid", adrenomedulin, C-terminal alpha-1 antitrypsin peptide)
- Female: 20 female adult patients after cardiac surgery. Drawing of patients blood for measurement of biomarkers ("penKid", adrenomedulin, C-terminal alpha-1 antitrypsin peptide) for AKI before and after cardiac surgery (times: 0, 6, 24, 72, 168 hours).
  Interventions: Diagnostic Test: Biomarker ("penKid", adrenomedulin, C-terminal alpha-1 antitrypsin peptide)

INTERVENTIONS:
Diagnostic Test: Biomarker ("penKid", adrenomedulin, C-terminal alpha-1 antitrypsin peptide) — Drawing of patients blood for measurement of biomarkers for AKI before and after cardiac surgery (times: 0, 6, 24, 72, 168 hours).

SUMMARY:
Acute kidney injury (AKI) is a common and major complication of cardiac surgery. The aim of this study is to evaluate the use of a fragment of proencephalin in plasma and other biomarkers as specific markers for early diagnosis of AKI and the need of renal replacement therapy after cardiac surgery.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) is an abrupt loss of kidney function and occurs in up to 5-40% of patients who undergo cardiac surgery; dialysis being required in approximately 2-15% of all patients. AKI is a common problem in critically ill patients and is independently from underlying diseases associated with increased morbidity and mortality (to progressive loss of kidney function, cardiovascular disease, and death). Unfortunately, chronic kidney disease is often overlooked in its earliest, most treatable stages. Implementation of novel biomarkers into the clinical practice that reliably identify patients at risk or at an early stage of AKI could offer more efficient management strategies may lead to better outcomes in critically ill patients.

Kidney disease usually progresses silently, often destroying most of the kidney function before causing any symptoms. AKI was defined using the Kidney Disease Improvement Global Outcome (KDIGO) definition. The standard key tests (increase of serum creatinine and urine output) are late parameters after significant kidney injury.

In this study 20 female and 20 male adult patients before and after cardiac surgery should be included. From all patients basic demographic data, pre-morbidity, vital parameters, blood parameters, urine output, Illness severity scores (APACHE-II, SOFA, GCS), drug levels, microbiological results will be recorded. The aim of this study is to evaluate the use of a fragment of proencephalin in plasma "penKID", Spingotec GmbH, Berlin, Germany) and other biomarkers (ADM: adrenomedulin, CAAP: C-terminal alpha-1 antitrypsin peptide) as specific markers for early diagnosis of AKI and the need of renal replacement therapy. Bio-ADM is a water-soluble peptide hormone with a molecular weight of about 6kDa released mainly by endothelial cells. Its biological function is the control of vasodilation, an important regulator of blood pressure and organ perfusion. This biomarker predicts and diagnoses endothelial dysfunctions. C-terminal alpha-1 antitrypsin peptide (CAAP) is a novel sepsis and renal injury biomarker with immunomodulatory function, especially in human neutrophils, which supports its role in the host response and pathophysiology of sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, at least 18 years old
* Ability to consent to the study by patient or legal representative
* Cardiac surgery with use of extracorporeal circulation (ECC)
* Bypass (> 2; ACB) or bypass + heart valve surgery
* Two or three heart-valve operation

Exclusion Criteria:

* Dialysis-dependent patients with chronic, end-stage renal failure
* Pre-existing renal replacement therapy
* Infused prognosis (expected death in ≤ 12 hours despite maximal therapy)
* Inability to consent of participation in the research project, of the patient or of the patients representative
* Aortic surgery
* Endocarditis
* (Only) partial sternotomy (eg. aortic valve surgery)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Gender Based: Yes — 20 female and 20 male patients.
Study Population: All patients undergoing cardiac surgery and fulfilling the inclusion criteria should be screened for the study at the university hospital of Rostock, Germany at one of the two different intensive care units PIT 1 and 2 at the Department of Anaesthesiology and Intensive Care or at the Department of Cardiac Surgery.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-07-27 (Actual); Primary Completion 2021-07 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
AKI 0 h | after operation (surgery): 0 hours
  Diagnosis and severity of acute kidney injury following the KDIGO-criteria
AKI 6 h | after operation (surgery): 6 hours
  Diagnosis and severity of acute kidney injury following the KDIGO-criteria

SECONDARY OUTCOMES:
SOFA | before operation, after operation (times: 0, 6, 24, 72 and 168 hours
  SOFA-Score

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sauer, MD, Principal Investigator — University Hospital of Rostock, Germany
Locations (1):
- Intensive Care Units PIT 1+2, University hospital Rostock, Rostock, Germany